CLINICAL TRIAL: NCT05685914
Title: Outcomes of Endoscopic Operation in COVID-19 Infection: Cohort Study.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Other Study IDs: qiwu
Record Dates: First submitted 2023-01-12; First posted 2023-01-17 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-01

CONDITIONS: COVID-19; Surgery-Complications
MeSH Terms: conditions — COVID-19 | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: endoscopic surgery — Emergency or elective surgery

SUMMARY:
The goal of this observational study is to determine 30-day mortality and post endoscopic surgery complications in patients with COVID-19 infection who undergo endoscopic surgery.This results will inform future risk stratification, decision making and improve patient's clinical care.This study is an investigator-led, non-commercial, non-interventional study is extremely low risk, or even zero risk.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing any type of endoscopic surgery in an operating theatre and these patients had COVID-19 infection either at the time of surgery or within 30 days of surgery.

Exclusion Criteria:

* If COVID-19 infection is diagnosed >30 days after discharge, the patient should not be included.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing endoscopic surgery done in an operating theatre by a surgeon.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-31 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  Death up to 30-days post surgery

SECONDARY OUTCOMES:
postoperative complications | 30 days
  Determine postoperative complications one month after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, China

IPD SHARING:
Plan to Share IPD: No